CLINICAL TRIAL: NCT04618445
Title: Prevalence of Temporomandibular Joint Disorders Among Egyptian University Undergraduate Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maram Ahmed Taema, Assistant Lecturer, Cairo University
Other Study IDs: 01112020
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: TMD; Bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Undergraduate students: prevalence of TMD among undergraduate students
  Interventions: Behavioral: some risk factors that might be correlated with TMD

INTERVENTIONS:
Behavioral: some risk factors that might be correlated with TMD — Fonesca questionnaire

SUMMARY:
This study will take place in Egypt. Undergraduate students from different faculties of the Egyptian Universities will participate. The study began in December 2020.

DETAILED DESCRIPTION:
Matching criteria and allocation ratio: The planned study a single arm cross sectional study, in which the prevalence of students of TMD will be reported. The association between TMD and other variables will be also studied. Therefore, no matching criteria or allocation ratio are required.

Variables It has been shown from literature that many variables are associated with TMD. It was therefore, decided to study the correlation between these variables with TMD among Egyptian population via a regression model once the assumption for regression analysis are satisfied. Binary variables are analyzed through logistic regression, while continuous data through a multivariable regression analysis. If one of the assumptions for regression analysis is violated, a subgroup analysis for each variable will be considered.

These Variables include gender, age, psychological stress, oral habits, parafunctional activities as gum chewing, previous dental treatments , previous trauma to jaws.

Data sources and management Data sources, the answered questionnaires and subsequent spread sheets will only be shared by the team members.

Addressing potential sources of bias Selection bias: an email will be sent to all the students through their university email addresses. Due to the COVID-19 situation only convenient sampling could be used. whenever possible printed questionnaires are handed to the students.

Quantitative variables: Handling of quantitative variables in the analyses None of the data is a continuous variable. All exposure factors are binary or categorical data. Therefore, no plans are set for simplifying continuous data or converting them into binary ones.

ELIGIBILITY:
Inclusion Criteria:

1. -Undergraduate students in Egyptian universities
2. Age ranges from 18-45 years
3. Males and females

Exclusion criteria

1. school students
2. students not living in egypt

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All undergraduate students in Egyptian Universities
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of TMDs in Egyptian university students | 3 months
  Fonseca Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ramsis Magdy, BDS, Principal Investigator — Cairo University; Azza Hussein, PhD, Study Chair — Cairo University; Iman Radi, PhD, Study Director — Cairo University; Maram Taema, Master, Study Director — Cairo University; Amr Nagib, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No